CLINICAL TRIAL: NCT04775732
Title: Ultra-proactive Therapeutic Drug Monitoring of Infliximab Based on Point-of-care-testing in Inflammatory Bowel Disease: a Pragmatic Trial
Brief Title: Ultra-proactive Therapeutic Drug Monitoring in Inflammatory Bowel Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imelda GI Clinical Research Center (Other)
Responsible Party: Principal Investigator, Peter Bossuyt, MD, Imelda GI Clinical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200840
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Crohn Disease; Ulcerative Colitis
Keywords: therapeutic drug monitoring; inflammatory bowel disease; point of care testing; infliximab
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: pragmatic cluster trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultra proactive arm (Experimental)
  Interventions: Biological: infliximab therapeutic drug monitoring
- reactive arm (Active Comparator)
  Interventions: Biological: infliximab therapeutic drug monitoring

INTERVENTIONS:
Biological: infliximab therapeutic drug monitoring — dose optimization of infliximab based on a predefined dosing algorithm

SUMMARY:
This is a comparative pragmatic trial in patients with UC and CD on maintenance treatment with IFX. All IBD patients from cohort A with maintenance IFX treatment at a referral IBD clinic are prospectively included between June and August 2018. An ultra-proactive IFX TDM algorithm is applied as follows. All patients have an ELISA TL measurement at baseline, of which the result determined the follow-up pathway: (A) TL between 3-7μg/mL: continuation at same dose and interval; (B) TL >7μg/mL: interval prolongation allowed; (C) TL <3μg/mL: interval shortening with minimum 2 weeks, with the next IFX TL measured using a POCT. (i) If the POCT showed an IFX TL <3μg/mL, dose was optimized ad hoc using a linear dosing formula (Dosen = (TL target * Dose n-1) / TL measured), followed by a new POCT test at next visit with the same interval. (ii) If the POCT showed an IFX TL ≥3µg/mL, no additional dose was given and routine TL testing with ELISA was retaken at next visit. At every visit this algorithm was reapplied to all patients.

The patients from cohort A will be compared with the patients from cohort B. The patients in cohort B receive maintenance IFX treatment at a referral IBD clinic during the same period. Dose adjustment are done based on standard of care reactive TDM of IFX and clinical symptoms. Data will be collected retrospectively to avoid treatment optimization bias.

ELIGIBILITY:
Inclusion Criteria:

* all adult IBD patients treated for at least 14 weeks with infliximab were included

Exclusion Criteria:

* induction treatment with infliximab (<14 weeks)
* treatment with other biological for IBD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
number of patients with infliximab failure | one year
  number of patients with infliximab failure after one year (infliximab failure = infliximab discontinuation, IBD related surgery, IBD related hospitalization, add-on IBD treatment, and allergic reaction to infliximab)

SECONDARY OUTCOMES:
number of TL measurements per patient per year | one year
percentage of interval changes (shortening, prolongation, bidirectional) | one year
number of patients with infliximab discontinuation | one year
  number of patients with discontinuation of infliximab
percentage of patients with sustained clinical remission | one year
  number of patients with physician global assessment <1 and all visits
number of patients with mucosal remission | one year
  number of patients with mucosal remission after one year. (Mucosal remission = simple endoscopic score for CD <3, Rutgeertscore <i2 for, Mayo endoscopic subscore <1 and faecal calprotectin <250 µg/ml. Endoscopy and/or faecal calprotectin between 6 and 12 months after inclusion. If endoscopy and faecal calprotectin at the same moment, then endoscopy was dominant)

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Imelda GI clinical research center, Bonheiden
  - AZ Sint Lucas, Ghent

IPD SHARING:
Plan to Share IPD: Undecided